CLINICAL TRIAL: NCT01140178
Title: A Phase la Trial of Photodynamic Therapy With HPPH (2-1 (Hexyloxyethyl)-2-devinylpyropheophorbide-a) for Treatment of Dysplasia, Carcinoma in Situ and T1 Carcinoma of the Oral Cavity and/or Oropharynx.
Brief Title: A Trial of Photodynamic Therapy With HPPH for Treatment of Dysplasia, Carcinoma in Situ and T1 Carcinoma of the Oral Cavity and/or Oropharynx
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 170910
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Dysplasia; Carcinoma of the Oral Cavity; Carcinoma of the Oropharynx
Keywords: Photodynamic Therapy; Oral dysplasia; oral cavity carcinoma; oropharynx carcinoma.
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HPPH (Experimental): a fixed HPPH dose of 4 mg/m2 infused over 1 hour, and 24 hours later light doses escalating from 100 J/cm2 to 125 and 140 J/cm2, respectively.
  Interventions: Drug: HPPH

INTERVENTIONS:
Drug: HPPH — Given IV

SUMMARY:
Recent literature suggests that certain patients with squamous cell cancers of the head and neck region may benefit from photodynamic therapy whether or not they may have received prior therapy, e.g. radiation therapy

DETAILED DESCRIPTION:
We propose to initiate a Phase 1 a clinical trial using HPPH and 665 nm light in patients with cancer of the oral cavity and/or oropharynx, including lesions of moderate to severe dysplasia, squamous carcinoma in situ and T1 squamous cells carcinoma. The study will employ a fixed HPPH dose of 4 mg/m2 infused over 1 hour, and 24 hours later light doses escalating from 100 J/cm2 to 125 and 140 J/cm2, respectively. The primary goal is the determination of the maximally tolerated PDT dose. Preliminary evidence for PDT efficacy wil also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe dysplasia and/or squamous carcinoma-in-situ of the oral cavity and/or oropharynx.
* Patients with T1 squamous cell carcinoma of the oral cavity and/or oropharynx.
* Patient may have primary and/or recurrent lesions to be treated.
* Diagnosis must confirmed by biopsy.
* Prior therapy of any type is allowed.
* Male or female patients at least 18 years old. Female patients must not be pregnant and must be practicing a medically acceptable form of birth control, be sterile or post-menopausal. Male patients should be using a medically acceptable form of birth control or be sterile.
* Patients must have an ECOG score of 0-2 (Appendix A 1 ).
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Patients with T2 or greater squamous cell carcinoma.
* True tongue base lesions (as determined by the treating physician).
* Patients with severe trismus that prevents adequate access to the lesion for treatment light delivery (as determined by the treating physician).
* Porphyria or hypersensitivity to porphyrin or porphyrin-like compounds.
* Patients with impaired hepatic (alkaline phosphatase (hepatic) or SGOT;:3 times the upper normal limits).
* Patients with minimal impairment of renal function (total serum bilirubin;: 2 mg/dl, serum creatinine;: 2 mg/dl)
* Unwilling or unable to follow protocol requirements.
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug and or light treatment.
* Patients on concurrent chemotherapy or radiation therapy or less than 4 weeks after the last dose of chemotherapy or radiation therapy.

Inclusion of Women and Minorities:

* Both men and women and members of all races and ethnic groups are eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-06-08 (Actual); Primary Completion 2013-01-29 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Toxicity | 6 weeks
  To determine the maximally tolerated dose in the oral cavity and/or oropharynx of photodynamic therapy (PDT) using HPPH (2-1 (hexyloxyethyl)-2- devinylpyropheophorbide-a) and 665 nm light.

SECONDARY OUTCOMES:
Tumor response | 3 months
Response of dysplasia, CiS and selected patients with T1 squamous cell carcinoma of the oral cavity and/or oropharynx using photodynamic therapy (PDT) with HPPH (2-1 (hexyloxyethyl)-2-devinylpyropheophorbide-a) and 665 nm light. | 3 months
Amount of HPPH in the blood prior to light treatment. | 3 months
Biomarkers, i.e. STAT3 crosslinks and/or activation status of pro-survival signaling molecules before and after PDT treatment. | 3 months
To determine non-invasively HPPH fluorescence and blood flow in To determine non-invasively HPPH fluorescence and blood flow in tumor and surrounding normal tissue before and after PDT | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Arshad, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States